CLINICAL TRIAL: NCT04352322
Title: Effectiveness of Oral Hyaluronic Acid (A+ HA(tm), TOP Pharm.) in Knee Osteoarthritis: Clinical Trial
Brief Title: Effectiveness of Oral Hyaluronic Acid in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: TOP Pharm & Medicalware (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR101-IRB2-033-1
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A+HA(tm) (Experimental): 20 ml oral solution of hyaluronic acid mixture in combination with glucosamine and chondroitin in a bottle. Administration with 250~500 ml water under fasting condition in the morning.
  Interventions: Dietary Supplement: A+HA(tm)
- Placebo (Placebo Comparator): 20 ml oral solution without active ingredients in a bottle. Administration with 250~500 ml water under fasting condition in the morning.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: A+HA(tm) — oral solution of hyaluronic acid mixture in combination with glucosamine and chondroitin
  Arms: A+HA(tm)
Dietary Supplement: Placebo — oral solution with no active ingredients
  Arms: Placebo

SUMMARY:
This study was a randomized, double-blind, placebo-controlled study evaluating the efficacy of an oral liquid HA supplement (A+HA) in symptoms relief and improvement of quality of life in knee osteoarthritis patients with mild knee pain.

DETAILED DESCRIPTION:
Subjects were initially screened at the Randomization/Baseline Visit (Week 0). Eligible subjects were randomized at the same visit into the treatment period and received the assigned treatment in a double-blind fashion for 8 weeks. During the 8 weeks treatment period, there were three follow-up visits requested (Week 2, Week 4 and Week 8). Efficacy was measured by using Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Short Form-36 (SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age >= 40 years old
* Diagnosed with knee OA which met the definition of Ahlbӓck classification12 and had knee joint symptoms within 30 days prior to enrollment

Exclusion Criteria:

* Had administered glucosamine one month prior to enrollment
* Had known allergy to oral HA
* BMI ≧40 kg/m2
* Knee OA was caused by occupational hazard or sports injury
* Patients with known other causes of arthritis (infectious rheumatoid or psoriatic arthritis), bony or soft tissue malignancy or peripheral neuropathy involving the lower extremities, cardiopulmonary disease which limited walking more than knee pain, knee instability defined as a report of knee buckling or locking within the past month of the study knee, major neurological deficit that affected gait, psychiatric illness that limited informed consent or Parkinsonism
* Women in pregnancy
* Wheel chair users

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
WOMAC | 8 weeks
  Mean change from baseline to 8 weeks. The higher the score, the greater the severity.

SECONDARY OUTCOMES:
SF-36 | 8 weeks
  Mean change from baseline to 8 weeks. A higher score indicates a better QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Shyu-Jye Wang, MD, Principal Investigator — China Medical University Hospital
Locations (1):
- TOP Pharm. & Medicalware, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang SJ, Wang YH, Huang LC. The effect of oral low molecular weight liquid hyaluronic acid combination with glucosamine and chondroitin on knee osteoarthritis patients with mild knee pain: An 8-week randomized double-blind placebo-controlled trial. Medicine (Baltimore). 2021 Feb 5;100(5):e24252. doi: 10.1097/MD.0000000000024252. PMID 33592868